CLINICAL TRIAL: NCT00473317
Title: Sunlight Exposures Effect on Serum Vitamin D Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Laura Armas, Creighton University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Creighton3
Record Dates: First submitted 2007-05-11; First posted 2007-05-15 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Vitamin D Deficiency
Keywords: sunlight; UVB; Vitamin D
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): All subjects in this study will be in the active arm
  Interventions: Behavioral: Sun Exposure

INTERVENTIONS:
Behavioral: Sun Exposure — Each subject will wear a swimming suit and be exposed to sunlight for 30 minutes total (15 minutes lying on back, 15 minutes lying on stomach).

SUMMARY:
When people eat a meal, some, but not all of the calcium in that meal is absorbed, that is, moved into the bloodstream. When the skin is exposed to sunlight during summer months, Vitamin D is made there and then modified into more active forms by the liver and kidneys. These more active forms of Vitamin D improve calcium absorption. Many adults living in the U.S. have little or no sun exposure and are low in Vitamin D. We know that specific wavelengths of sunlight called Ultraviolet-B cause Vitamin D to be made in the skin.

DETAILED DESCRIPTION:
At the beginning of the study we will measure your height, weight, skin color, and draw blood to measure your blood levels of Vitamin D and 25-hydroxyvitamin D. Each subject will wear a swimming suit and be exposed to sunlight for 30 minutes total (15 minutes lying on back, 15 minutes lying on stomach).We will draw blood for Vitamin D and 25-hydroxyvitamin D on days 1,2,3,5, and 7 after sunlight exposure. There will be six blood draws for a total of 102 cc of blood drawn (about 3 ½ teaspoons drawn each time).

ELIGIBILITY:
Inclusion Criteria:

* healthy males or females ages19-50 with "light" skin (self-assessed as Fitzpatrick skin type I-III) with minimal sun exposure and exogenous sources of vitamin D.

Exclusion Criteria:

* less than 16 oz milk per day, less than 10 hours of sun per week, no Vitamin D supplements, no anticonvulsants, no barbiturates, no steroids, no meds that increase photosensitivity, no granulomatous disease, no liver or kidney disease, no history of skin cancer, and BMI less than 30.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2007-07; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The goal of this study is to correlate vitamin D response and 25(OH)D response to sun exposure with most of the body (90 %) exposed to 0.25 hour of July sunlight at 41.2º N latitude and at approximately 1-2 pm in the afternoon. | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Armas, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States